CLINICAL TRIAL: NCT06723808
Title: Relationship Between Leisure-Time Physical Activity and Work Ability in University Staff With Different Occupational Demands: A Cross-Sectional Study With a Gender Perspective
Brief Title: Physical Activity and Work Ability in University Staff
Status: Recruiting | Type: Observational
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Laura Lorenzo Gallego, University Professor and Director of Physiotherapy in Women's Health Research Group, University of Alcala
Other Study IDs: CEID/2024/3/061
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-11

CONDITIONS: Work Ability
Keywords: Physical Activity; Working Conditions; Recreational Activities; Sedentary Behavior; Gender Perspective
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- University staff in the Autonomous Community of Madrid: This cohort consists of university staff from the University of Alcalá, including both men and women, with varying occupational physical activity (OPA) levels.
  Interventions: Other: Leisure-Time Physical Activity and Occupational Physical Activity

INTERVENTIONS:
Other: Leisure-Time Physical Activity and Occupational Physical Activity — This study does not involve a specific intervention but explores the relationship between leisure-time physical activity (LTPA) and occupational physical activity (OPA) in university staff, with a focus on work ability, musculoskeletal disorders, and quality of life.

SUMMARY:
The goal of this observational study is to explore the relationship between leisure-time physical activity (LTPA) and work ability in university staff, with a focus on occupational physical activity (OPA) and gender. The main question it aims to answer is:

How does leisure-time physical activity (LTPA) influence work ability in university staff, considering their occupational physical activity (OPA) and gender?

Participants from the University of Alcalá will complete an online survey, which includes sociodemographic data and validated questionnaires on LTPA, OPA, work ability, musculoskeletal disorders, health-related quality of life, and workload.

DETAILED DESCRIPTION:
Introduction: 39.17% of the population in the Autonomous Community of Madrid (CAM) does not meet the physical activity recommendations set by the World Health Organization, representing a significant public health issue and considerable socioeconomic costs. Sex, gender, and working conditions are key determinants of leisure-time physical activity (LTPA). However, there are few studies aimed at understanding these sociocultural barriers.

Objective: To describe the association between LTPA and work ability, depending on occupational physical activity (OPA), among university staff in CAM, with a gender perspective. Secondly, to describe the relationship between the prevalence of musculoskeletal disorders at work, health-related quality of life (HRQoL), physical and mental workload, functional capacity, and working conditions with the aforementioned association.

Methodology: Cross-sectional descriptive study. The study population will consist of a representative sample of 885 workers from the University of Alcalá (Alcalá de Henares, Madrid), selected by snowball non-probability sampling. Participants will complete an ad hoc form (Microsoft Forms) including sociodemographic data (working hours, type of service, main task, income, menopause, etc.) and validated questionnaires in Spanish. The variables collected through these questionnaires will include LTPA and OPA (Global Physical Activity Questionnaire), work ability (Work Ability Index), prevalence of musculoskeletal disorders at work (Nordic Musculoskeletal Questionnaire), HRQoL (SF-12), and physical and mental workload (NASA Task Load Index).

Discussion: Improving understanding of the social determinants of physical activity in this population could facilitate the design of culturally sensitive interventions, thus making them more effective in reducing the economic and health costs of sedentary behavior.

ELIGIBILITY:
Inclusion Criteria:

* University staff from different departments of the University of Alcalá who are able to understand Spanish.

Exclusion Criteria:

* Individuals with cognitive limitations that hinder their ability to comprehend information, respond to questionnaires, or consent to participation in the study.
* Individuals with neurological impairments or a diagnosis of severe mental illness.
* Individuals with uncontrolled cardiorespiratory diseases or diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include staff members from the University of Alcalá, specifically those belonging to the PDI (teaching and research staff) and PTGAS (administrative and service staff) categories. Participants will be selected from various departments within the university. The population will consist of employees who are able to understand Spanish and who meet the inclusion criteria for the study, focusing on those with a range of job roles and occupational demands. This diverse group allows for an examination of the relationship between physical activity, work ability, and other health-related variables across different occupational contexts within the university setting.
Sampling Method: Non-Probability Sample
Enrollment: 876 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Leisure-Time Physical Activity (LTPA) | At the same time as the recruitment
  Leisure-time physical activity refers to any physical activity performed during free time, not related to work or mandatory responsibilities. This includes activities such as walking, jogging, cycling, sports, or any form of exercise done for enjoyment, health, or fitness outside of regular occupational or household duties. LTPA is measured through Global Physical Activity Questionnaire (World Health Organization, 2001) that assess the frequency, duration, and intensity of activities performed during leisure time. It is an important determinant of overall health and well-being, with potential impacts on physical fitness, mental health, and work ability.
Occupational Physical Activity (OPA) | At the same time as the recruitment
  Occupational physical activity refers to the physical activity performed as part of an individual's job or work-related tasks. This includes movements such as walking, lifting, carrying, standing, or any other physical effort required by the nature of the work. OPA varies depending on the type of occupation, ranging from sedentary jobs with minimal physical exertion to physically demanding jobs that involve heavy lifting or manual labor. OPA is going to be assessed through Global Physical Activity Questionnaire (World Health Organization, 2001). It is an important factor influencing overall physical health, musculoskeletal health, and work ability. Understanding OPA can help identify how job-related physical activity influences worker well-being and performance.
Work Ability | At the same time as the recruitment
  Work ability refers to an individual's capacity to perform their job tasks effectively, considering their physical and mental health, skills, and work demands. It reflects how well a person's health and functional capacity match the requirements of their work. Work ability is influenced by various factors, including physical fitness, mental well-being, work environment, and personal characteristics such as age and job experience. In this study, work ability will be measured using the Work Ability Index (WAI), a validated questionnaire developed by the Finnish Institute of Occupational Health. The WAI assesses work ability through a series of questions related to perceived health, job demands, and the impact of health on work performance.

SECONDARY OUTCOMES:
Prevalence of Musculoskeletal Disorders and Work-Related and Daily Activity Injuries | At the same time as the recruitment
  This variable refers to the frequency of musculoskeletal disorders (MSDs) and injuries related to work activities and daily life. MSDs are conditions that affect the muscles, bones, joints, tendons, and ligaments, often leading to pain and disability. These disorders can be caused or aggravated by repetitive movements, poor ergonomics, or physical strain in both occupational and non-occupational contexts. The Nordic Musculoskeletal Questionnaire (NMQ) will be used to assess the prevalence of these disorders, as well as injuries related to work and daily activities. The NMQ is a widely used tool for identifying and evaluating musculoskeletal symptoms in different body regions. In this study, the questionnaire will be adapted to the Spanish population, following the methodology proposed by Gómez-Rodríguez et al. (2020).
Physical and Mental Workload | At the same time as the recruitment
  Physical and mental workload refers to the level of physical and cognitive effort required to perform a task or job. Physical workload includes factors such as physical exertion, body movements, and posture, while mental workload relates to cognitive demands, stress, and mental concentration required by the job. Both components contribute to the overall strain experienced by workers and can affect job performance, health, and well-being. The NASA Task Load Index (NASA-TLX) will be used to assess the physical and mental workload in this study. The NASA-TLX is a validated method developed by the National Aeronautics and Space Administration (NASA) to evaluate workload across multiple dimensions, including mental demand, physical demand, temporal demand, performance, effort, and frustration. This tool helps to quantify the subjective workload experienced by participants in various work scenarios.
Health-Related Quality of Life (HRQoL) | At the same time as the recruitment
  Health-related quality of life refers to an individual's overall well-being in relation to their health, encompassing both physical and mental health components. It evaluates how health conditions, including physical ailments and mental health issues, affect daily functioning, social interactions, and overall life satisfaction. In this study, HRQoL will be measured using the SF-12 Health Survey, a short form of the widely used SF-36 questionnaire. The SF-12 assesses 12 questions related to physical and mental health, covering areas such as physical functioning, role limitations due to physical or emotional problems, social functioning, and general health perceptions. This tool has been validated in various populations, including Spanish-speaking communities (Alonso, 1996).

OTHER OUTCOMES:
Sociodemographic Data | At the same time as the recruitment
  Age, sex, gender, BMI, place of residence, specific occupation, educational level, working hours, type of work shift, anthropometric characteristics, and, for women, whether they have entered menopause and since when. Optionally, marital status, annual income, and household tasks will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: María Torres Lacomba, PhD, MSc, PT, Study Director — University of Alcala. Phsyiotherapy in women's health research group.; Beatriz Navarro Brazález, PhD, MSc, PT, Study Director — University of Alcala. Phsyiotherapy in women's health research group.
Locations (2):
- Spain (2):
  - University of Alcala, Alcalá de Henares, Madrid
  - Faculty of Medicine and Health Sciences. University of Alcalá, Alcalá de Henares, Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lorenzo-Gallego L, Munoz-Pastor S, Menendez-Calvo MR, Navarro-Brazalez B, Torres-Lacomba M. Understanding the Link Between Physical Activity and Work Ability in University Staff: Protocol for a Gender-Sensitive Cross-Sectional Study. JMIR Res Protoc. 2025 Aug 28;14:e80298. doi: 10.2196/80298. PMID 40875988